CLINICAL TRIAL: NCT04121923
Title: Validation of a Novel Device for Screening Patients With Symptoms of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belun Technology Company Limited (Other)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PR 2018-259
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participant (Experimental): All patients scheduled for attended overnight in-lab polysomnography (PSG) will undergo PSG testing. On the same night of the PSG testing, these same patients will also wear the Belun Ring device. After the study, we will compare results of the Belun Ring device with the results of the PSG on the same patient. There will be no separate arm to test a different device.
  Interventions: Device: Belun Ring Pulse Oximeter

INTERVENTIONS:
Device: Belun Ring Pulse Oximeter — Belun Ring Pulse Oximeter allows measurement and analysis of oximetry, pulse rate, photo-plethysmography (PPG), and accelerometer signals from the proximal phalanx of index finger. Total sleep time (Ring-TST) and respiratory event index (Ring-REI) are estimated

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of the Belun Ring Pulse Oximetry system for screening of obstructive sleep apnea (OSA) in adults during standard polysomnography sleep study conditions. The primary outcome metric is the Apnea-Hypopnea Index (AHI).

The goal, in its entirety, is to evaluate the performance of the Belun Ring Pulse Oximeter during a standard polysomnography sleep study and its ability to compare to the determined Apnea-Hypopnea Index (AHI) of the subjects. It is expected that the Belun Ring Pulse Oximeter will adequately record SpO2, pulse rate, body position and heart rate variability throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent.
* Subject is 18 to 90 years of age.
* Subject must be willing and able to comply with study procedures and duration.
* Male or female of any race.

Exclusion Criteria:

* Subject requires oxygen therapy or noninvasive ventilation.
* Subject has a current diagnosis of chronic obstructive pulmonary disorder (COPD), neuromuscular disease, periodic limb movement, or narcolepsy.
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Subject is on medication known to interfere with heart rate, such as beta blockers, digoxin, or calcium receptor agonists.
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported).
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, which should be considered.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 2 years
  To evaluate the ability of the Belun ring pulse oximeter to correctly gauge the Apnea-Hypopnea Index (AHI).

CONTACTS AND LOCATIONS:
Locations (1):
- Mountain Sleep Diagnostics, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gu W, Leung L, Kwok KC, Wu IC, Folz RJ, Chiang AA. Belun Ring Platform: a novel home sleep apnea testing system for assessment of obstructive sleep apnea. J Clin Sleep Med. 2020 Sep 15;16(9):1611-1617. doi: 10.5664/jcsm.8592. PMID 32464087